CLINICAL TRIAL: NCT01534286
Title: A Randomized Double-Blind Placebo Controlled Trial to Determine the Status of Post Knee Chondroplasty Patients Administered Theramine Versus Placebo in Addition to Post Surgery Analgesics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit patients
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0201302
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Knee Pain; Knee Chondroplasty
Keywords: Prescription Medical Food; Theramine; Knee surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theramine (Active Comparator): Theramine 2 capsules three times per day in addition to post surgical analgesic medication.
  Interventions: Drug: Theramine
- Theramine-like Placebo (Placebo Comparator): Theramine-like placebo 2 capsules three times per day in addition to post surgical analgesic medication.
  Interventions: Drug: Theramine- like placebo

INTERVENTIONS:
Drug: Theramine — Theramine 2 capsules 3 times per day
  Arms: Theramine
Drug: Theramine- like placebo — Theramine-like placebo capsules 2 three times daily
  Arms: Theramine-like Placebo

SUMMARY:
The purpose of this study will be to show the patient response to analgesics taken post surgery when taken in combination with Theramine as opposed to Theramine-like placebo. The data collected will be used to show that patients have a shorter and lower post operative pain measurement and the time to discontinuation of analgesics is less in the active comparator group.

DETAILED DESCRIPTION:
No other decription

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed knee pain requiring chondroplasty knee arthroscopic surgery.
* Men and non-pregnant, non-lactating women over the age of 18 and under the age of 75, able to read, understand and sign English-language informed consent.
* If using psychoactive medication which might have analgesic effects, (i.e. anti-depressants or anti-consultants), treatment must be stable for at least three (3) months prior to study.
* For men and women of child-bearing potential, must be willing to use adequate contraception and not be pregnant or impregnate their partner during the entire time of study.
* Must be willing to commit to all clinical visits during study-related procedures.
* Require use of narcotics for pain relief.

Exclusion Criteria:

* Patients with significant neurologic impairment, as diagnosed on screening physical examination.
* Patients not fluent in English.
* Patients currently involved in a Workman's Compensation case related to this procedure.
* Receipt of an oral intramuscular or soft-tissue injection of corticosteroid within one (1) month prior to screening.
* History of substance abuse.
* History of malignancy, other than basal or squamous cell of the skin within the last 5 years.
* Tibial plateau fracture within 6 months prior to surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dose reduction of analgesic. | 28 days
  The primary efficacy outcome will be the overall dose reduction of analgesic in the Theramine active group versus the Theramine placebo group.

SECONDARY OUTCOMES:
Change in Visual Analogue Scale Evaluation (VASE) | 28 days
Change in second Knee pain scale. | 28 Days
Time to discontinuation of analgesic. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory V. Hickman, MD, Principal Investigator — Andrews-Paulos Research & Education Institute
Locations (1):
- Andrews-Paulos Research & Education Institute, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Too small data set to draw any conclusions

REFERENCES:
- See also: Related Info — http://tmedpharma.com